CLINICAL TRIAL: NCT03099226
Title: A Double-blind, Randomised, Placebo-controlled Study to Evaluate the Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Dose Regimens of Etamicastat (BIA 5-453) in Hypertensive Subjects
Brief Title: Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Dose Regimens of BIA 5-453
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-5453-201HT
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — etamicastat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - BIA 5-453 50 mg or placebo (Experimental): This study investigated the doses of 50, 100 and 200 mg of Etamicastat (BIA 5-453) during 10 days administered q.d. in the morning under fasting conditions.
  On Day 1 and Day 10, patients remained fasted from a minimum of 8 hours before drug administration until after the collection of the 4 hour PK timepoint. Individuals were served a meal following the 4 hour timepoint and had free access to a maximum of 2.5 litres of water per day. However they were not allowed to drink 1 hour before and 1 hour after the dosing except for the 250 mL taken with the IMP at administration.
  On other administrations days, patients remained fasted for a minimum of 8 hours before drug administration and the treatments were administered one hour before a standardized breakfast.
  The patients were administered between 7:00 and 9:00 o'clock a.m
  Interventions: Drug: Placebo; Drug: BIA 5-453
- Group 2 - BIA 5-453 100 mg or placebo (Experimental): This study investigated the doses of 50, 100 and 200 mg of Etamicastat (BIA 5-453) during 10 days administered q.d. in the morning under fasting conditions.
  On Day 1 and Day 10, patients remained fasted from a minimum of 8 hours before drug administration until after the collection of the 4 hour PK timepoint. Individuals were served a meal following the 4 hour timepoint and had free access to a maximum of 2.5 litres of water per day. However they were not allowed to drink 1 hour before and 1 hour after the dosing except for the 250 mL taken with the IMP at administration.
  On other administrations days, patients remained fasted for a minimum of 8 hours before drug administration and the treatments were administered one hour before a standardized breakfast.
  The patients were administered between 7:00 and 9:00 o'clock a.m
  Interventions: Drug: Placebo; Drug: BIA 5-453
- Group 3 - BIA 5-453 200 mg or placebo (Experimental): This study investigated the doses of 50, 100 and 200 mg of Etamicastat (BIA 5-453) during 10 days administered q.d. in the morning under fasting conditions.
  On Day 1 and Day 10, patients remained fasted from a minimum of 8 hours before drug administration until after the collection of the 4 hour PK timepoint. Individuals were served a meal following the 4 hour timepoint and had free access to a maximum of 2.5 litres of water per day. However they were not allowed to drink 1 hour before and 1 hour after the dosing except for the 250 mL taken with the IMP at administration.
  On other administrations days, patients remained fasted for a minimum of 8 hours before drug administration and the treatments were administered one hour before a standardized breakfast.
  The patients were administered between 7:00 and 9:00 o'clock a.m
  Interventions: Drug: BIA 5-453

INTERVENTIONS:
Drug: Placebo — Placebo blue hard gelatine capsules
  Arms: Group 1 - BIA 5-453 50 mg or placebo; Group 2 - BIA 5-453 100 mg or placebo
Drug: BIA 5-453 — Etamicastat (BIA 5-453) blue hard gelatine capsules - 50 Strength (mg)
  Other Names: Etamicastat

SUMMARY:
The purpose of this study was to characterise the plasma and urine pharmacokinetic profile of Etamicastat (BIA 5-453) and its metabolites after three multiple rising dose regimens of Etamicastat (BIA 5-453).

DETAILED DESCRIPTION:
Single centre, double-blind, randomised, placebo-controlled study of three dosage regimens of Etamicastat (BIA 5-453) in 3 groups of 8 hypertensive patients.

In each group, the study consisted of a 10-day multiple-dose period. Progression to the next dose level only occurred if the previous dose level was considered to be safe and well tolerated. An appropriate interval separated the investigation of doses to permit a timely review and evaluation of safety data prior to proceeding to a higher dose level.

ELIGIBILITY:
Inclusion Criteria:

1. A signed and dated informed consent form before any study-specific screening procedure is performed.
2. Male patients aged between 18 and 65 years (inclusive)
3. Body mass index (BMI) between 18 and 35 kg/m2 (inclusive)
4. Patients with essential hypertension, without previous treatment (but in which treatment was justified), defined at the selection visit as blood pressure (BP) after 10 minutes of rest in supine position of

   * diastolic blood pressure (DBP) ≥ 90 mmHg and/or,
   * systolic blood pressure (SBP) ≥ 140 mmHg
5. Patients with essential hypertension, with previous treatment, defined at the end of the screening period (i.e. after 3 weeks wash-out of antihypertensive treatment(s) and before D-1) as blood pressure (BP) after 10 minutes of rest in supine position of

   * diastolic blood pressure (DBP) ≥ 90 mmHg and/or,
   * systolic blood pressure (SBP) ≥ 140 mmHg
6. Naive or patients taking any class of antihypertensive treatment including (but not limited to) one of the following authorised treatments: B-blockers, diuretics, angiotensin-converting enzyme inhibitor (ACEI), angiotensin receptor blocker (ARB), calcium channel blockers. Patients observed a wash-out for their antihypertensive treatments of approximately 3 weeks.
7. Laboratory tests within the normal range of the laboratory (haematology, biochemistry and urinalysis) or considered as not clinically significant by the investigator.
8. Electrocardiogram recording on a 12-lead ECG without any clinically significant abnormality
9. Covered by National Health Insurance
10. Once clinical eligibility had been established, patients conducted 24 h ambulatory blood pressure monitoring (ABPM) at the end of the screening period, and after treatment wash-out for patients already treated. They had to meet the following off-treatment criteria for mean 24 h ambulatory blood pressure measurements to be included in the study:

    * Average daytime ambulatory systolic/diastolic BP ≥ 135 / 85 mm Hg and/or
    * Ambulatory night-time systolic/diastolic BP ≥ 120 / 70 mm Hg.

Exclusion Criteria:

Criteria associated with hypertension, associated risk factors, and target organ damage:

1. Severe hypertension (SBP≥180 mm Hg and/or DBP≥110 mm Hg) at any time during the study from screening period to end of study visit or in the medical history, malignant hypertension
2. Secondary hypertension (including known renovascular hypertension, pheochromocytoma)
3. Any recent history of coronary artery disease (in the previous 6 months) and including myocardial infarction, or precordial pain suggesting angina pectoris and coronary revascularisation
4. Any recent history of cardiac failure (in the previous 6 months)
5. Any recent history of cerebrovascular stroke or transient ischemia (in the previous 6 months)
6. Any known aortic or mitral valve stenosis or hypertrophic obstructive myocardiopathy
7. Any known severe ocular complication of hypertension (stage III or IV retinopathy),
8. Any history of ventricular rhythm disorders (torsades de pointes, ventricular tachycardia, polymorphic ventricular extra-systoles except isolated extra-systoles), auricular disorders (fibrillation or flutter).
9. Any surgical or medical condition that might significantly alter the absorption, distribution, metabolism, or excretion of Etamicastat (BIA 5-453)
10. Presence or history of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, haematological, neurological or psychiatric disease.
11. Frequent headaches and/or migraine, recurrent nausea and/or vomiting (more than twice a month).

    Criteria associated with patient characteristic:
12. History or presence of drug dependence.
13. Patients smoking more than 10 cigarettes per day
14. History of alcoholism within 1 year before day 1. Consumption of more than 50 g of ethanol per day (12.5 cL glass of 10° [10%] wine = 12 g; 4 cL of aperitif, 42° [42%] whiskey = 17 g; 25 cL glass of 3° [3%] beer = 7.5 g; 25 cL glass of 6° [6%] beer = 15 g
15. Participation in a drug trial within 3 months preceding the selection visit.
16. Positive result from the hepatitis serology for hepatitis B (HBs Ag) and/or hepatitis C (HCV Ab).
17. Positive result for HIV1+2 serology.
18. Positive Urine Drug Screen (UDS) (amphetamines, benzodiazepines, ecstasy, cocaine, opiates).
19. Loss of greater than 400 mL or blood donation within the last 3 months.

    Criteria associated with concomitant diseases:
20. Patients taking one of the following treatments: aldosterone antagonists, nitrite derivatives.
21. Presence or history of any allergic or unusual reaction to drugs.
22. Excessive consumption of beverages containing xanthine bases (more than six cups or glasses per day) or inability to stop consumption during the hospitalization.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-07-15 (Actual); Primary Completion 2009-04-03 (Actual); Study Completion 2009-04-03 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum observed plasma concentration (Plasma results on Day 1) | D1 pre-dose, and H0.5 , 1, 2, 3, 4, 5, 6, 8, 10, 12, 16 post-dose
  Plasma pharmacokinetic parameters (SD) following single and repeated doses of 50, 100, and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects
tmax: time to reach maximum plasma concentration (Plasma results on Day 1) | D1 pre-dose, and H0.5 , 1, 2, 3, 4, 5, 6, 8, 10, 12, 16 post-dose
  Plasma pharmacokinetic parameters (SD) following single and repeated doses of 50, 100, and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects
AUC0-t: Area under the plasma concentration-time curve from time zero to last measurable plasma concentration (Plasma results on Day 1) | D1 pre-dose, and H0.5 , 1, 2, 3, 4, 5, 6, 8, 10, 12, 16 post-dose
  Plasma pharmacokinetic parameters (SD) following single and repeated doses of 50, 100, and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects
AUC0-24: AUC from time zero to 24h-post dose (Plasma results on Day 1) | D1 pre-dose, and H0.5 , 1, 2, 3, 4, 5, 6, 8, 10, 12, 16 post-dose
  Plasma pharmacokinetic parameters (SD) following single and repeated doses of 50, 100, and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects
Cmax: Maximum observed plasma concentration (Plasma results on Day 10) | D10 pre-dose, and H0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12,16, 24, 48 and 72 h post-dose
  Plasma pharmacokinetic parameters (SD) following single and repeated doses of 50, 100, and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects
tmax: time to reach maximum plasma concentration (Plasma results on Day 10) | D10 pre-dose, and H0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12,16, 24, 48 and 72 h post-dose
  Plasma pharmacokinetic parameters (SD) following single and repeated doses of 50, 100, and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects
AUC0-t: Area under the plasma concentration-time curve from time zero to last measurable plasma concentration (Plasma results on Day 10) | D10 pre-dose, and H0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12,16, 24, 48 and 72 h post-dose
  Plasma pharmacokinetic parameters (SD) following single and repeated doses of 50, 100, and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects
AUC0-24: AUC from time zero to 24h-post dose (Plasma results on Day 10) | D10 pre-dose, and H0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12,16, 24, 48 and 72 h post-dose
  Plasma pharmacokinetic parameters (SD) following single and repeated doses of 50, 100, and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects
C max : Maximum excretion rate (Urine results on Day 1) | D1 pre-dose, and 0-4, 4-8, 8-12, 12-24 h post-dose
  Urine pharmacokinetic parameters (SD) following single and repeated doses of 100 and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects
tmax : Time of Maximum Excretion Rate (Urine results on Day 1) | D1 pre-dose, and 0-4, 4-8, 8-12, 12-24 h post-dose
  Urine pharmacokinetic parameters (SD) following single and repeated doses of 100 and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects
AURC(0-tlast) : Area Under the Urine Excretion Curve from time zero to last time (Urine results on Day 1) | D1 pre-dose, and 0-4, 4-8, 8-12, 12-24 h post-dose
  Urine pharmacokinetic parameters (SD) following single and repeated doses of 100 and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects
AmtCUM : Cumulative Amount of Drug excreted in urine (Urine results on Day 1) | D1 pre-dose, and 0-4, 4-8, 8-12, 12-24 h post-dose
  Urine pharmacokinetic parameters (SD) following single and repeated doses of 100 and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects
C max : Maximum excretion rate (Urine results on Day 10) | D10 pre-dose, and 0-4, 4-8, 8-12, 12-24, 24-48, 48 72 h post-dose
  Urine pharmacokinetic parameters (SD) following single and repeated doses of 100 and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects
tmax : Time of Maximum Excretion Rate (Urine results on Day 10) | D10 pre-dose, and 0-4, 4-8, 8-12, 12-24, 24-48, 48 72 h post-dose
  Urine pharmacokinetic parameters (SD) following single and repeated doses of 100 and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects
AURC(0-tlast) : Area Under the Urine Excretion Curve from time zero to last time (Urine results on Day 10) | D10 pre-dose, and 0-4, 4-8, 8-12, 12-24, 24-48, 48 72 h post-dose
  Urine pharmacokinetic parameters (SD) following single and repeated doses of 100 and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects
AmtCUM : Cumulative Amount of Drug excreted in urine (Urine results on Day 10) | D10 pre-dose, and 0-4, 4-8, 8-12, 12-24, 24-48, 48 72 h post-dose
  Urine pharmacokinetic parameters (SD) following single and repeated doses of 100 and 200 mg of Etamicastat (BIA 5-453) in hypertensive subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided